CLINICAL TRIAL: NCT02683902
Title: The Effect of Hypocaloric Diet Associated With tDCS on Weight Loss and Metabolic Profile: a Pilot, Double Blind, Randomized, Placebo-controlled Study
Brief Title: The Effect of Hypocaloric Diet Associated With tDCS on Weight Loss and Metabolic Profile
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-0119
Record Dates: First submitted 2016-01-11; First posted 2016-02-17 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-08

CONDITIONS: Prediabetes; Obesity; Weight Loss; Diabetes; Overweight
Keywords: prediabetes; tDCS; transcranial direct current stimulation; obesity; diabetes
MeSH Terms: conditions — Prediabetic State; Obesity; Weight Loss; Diabetes Mellitus; Overweight | interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tDCS + Diet (Active Comparator): The participants will receive active tDCS treatment every day for 5 days per week, a total of 20 sessions. They will also be prescribed a hypocaloric dietary during these 4-week treatment.
  Interventions: Device: Active tDCS; Behavioral: Hypocaloric diet
- Sham tDCS + Diet (Sham Comparator): The participants will receive sham tDCS treatment every day for 5 days per week, a total of 20 sessions. They will also be prescribed a hypocaloric dietary during these 4-week treatment.
  Interventions: Behavioral: Hypocaloric diet; Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — The anode electrode will be placed over F4 position and the cathode electrode over F3, right and left respectively (using EEG 10/20 system). The electric current will be ramped up until it reaches 2 milliampere (mA), and subjects will be stimulated for 20 min.
  Other Names: Active
  Arms: Active tDCS + Diet
Behavioral: Hypocaloric diet — A hypocaloric dietary prescription and individual counseling from a dietician in order to reduce 3% of their initial weight over 4-week treatment.
  Other Names: Diet
Device: Sham tDCS — The electrodes will be placed at the same positions as in active stimulation; however, the device will be turned off after 30 s of stimulation.
  Other Names: Placebo
  Arms: Sham tDCS + Diet

SUMMARY:
To compare four weeks of transcranial direct current stimulation (tDCS) versus placebo associated with a reduced caloric diet on weight loss, glycemic control and regulators of hunger and satiety in overweight or obese subjects with different degrees of glucose tolerance, submitted to hypocaloric diet.

DETAILED DESCRIPTION:
In order to assess whether tDCS treatment associated with a reduced caloric diet can improve weight loss, overweight or obese subjects will be recruited by advertisement on the web page of Porto Alegre Clinical Hospital, local newspaper and television, or referred by a doctor or nutritionist, from external to HCPA services. After screening and selection, patients will undergo a clinical, laboratory and nutritional evaluation. There will be a standard assessment protocol that includes: a complete clinical evaluation and socioeconomic status, assessment of physical activity, questionnaires of quality of life, sleep, depression and anxiety and body composition assessment.

In the laboratory evaluation the biochemistry exams include an oral glucose tolerance test (OGGT 75g), a meal tolerance test (MTT), serum glucose, Cholesterol, HDL-cholesterol, triglycerides, glycated hemoglobin and glycated albumin. The resting metabolic rate will be determine by indirect calorimetry. Besides, a 100-mm visual-analog scales will be used to measure a self-reported ratings of appetite, hunger, satiety and food craving.

Patients will also be prescribed a low caloric diet and individual counseling from a dietician in order to reduce 3% of their initial weight over 4-week treatment. Moreover, they will do one tDCS session a day (active or sham stimulation as previous randomization) for 5 consecutive days, during these four weeks of treatment (20 sessions).

Transcranial direct current stimulation (tDCS) is a non-invasive method of brain stimulation in which a small current is applied to the scalp. This technique uses a weak safety current of 2 milliampere (mA) for 20 minutes which may increase (anodal tDCS) or decrease (cathodal tDCS) cortical excitability.

During all of tDCS sessions, a film with images of food that usually elicit craving will be presented and after the end of each session, visual analog scales will be applied to assess hunger, satiety and presence of food craving. Finally, attention and mood scales will be applied periodically in addition to a questionnaire of adverse effects and use of tDCS.

At the end of the 4-week diet and tDCS, all patients will be submitted to the same clinical, laboratory, nutrition and feeding behavior exams applied at baseline.

Finally, participants should come in 3 and 6 months after the end of the protocol for reassessment weight, body composition by bioelectrical impedance and answer questionnaires.

An interim analysis will be performed when 12 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

1. Women of childbearing potential who are using medically approved birth control methods (eg hormonal contraceptives, intra uterine device (IUDs), barrier contraception) and who agree to use the same methods of contraception throughout the course of the study.
2. BMI 25 ≥ 35 Kg/m2 at screening
3. Stable weight for at least 12 weeks prior to screening
4. Able and willing to provide written informed consent and to comply with the requirements of the study protocol

Exclusion Criteria:

1. Pregnant or intend to become pregnant during the study period or who are currently breastfeeding.
2. Women in perimenopause / menopause, or postmenopausal status, or who have had early menopause (under 40 years) or have had a hysterectomy or oophorectomy.
3. Diagnosis or history of diabetes Mellitus type 1, diabetes resulting from pancreatic injury or secondary forms of diabetes, such as, for example, Cushing's syndrome and acromegaly.

   3.1. Metabolic and acute complications of diabetes such as ketoacidosis and hyperosmolar coma within the past six months.
4. Gastrointestinal disease clinically symptomatic including, among others, inflammatory bowel disease and/or malabsorption diseases.
5. Have received nutritional counseling in the last six months by a nutritionist.
6. History of severe depression or other serious psychiatric comorbidities.
7. History of gastric bypass, antrectomy or small bowel resection.
8. History of chronic pancreatitis or idiopathic acute pancreatitis
9. Myocardial infarction (MI), coronary arteries bypass surgery, post-transplant cardiomyopathy or stroke in the last 6 months
10. Any abnormality in clinical laboratory tests which might prevent safe participation in the study
11. Diagnosed and / or treated tumor (except basal cell skin cancer, carcinoma in situ of the cervix or prostate cancer in situ) in the last five years.
12. History of known hemoglobinopathy and chronic anemia.
13. Donation of one unit (500 ml) of blood or more, significant blood loss equivalent to at least one unit of blood within the last 2 weeks or blood transfusion in the past 8 weeks.
14. Treatment with any oral antidiabetic drugs and / or herbal preparations or medications that do not require a prescription and can affect glycemic control within 12 weeks prior to screening.
15. Chronic treatment with oral or parenteral corticosteroids (> 7 consecutive days of treatment) within 4 weeks prior to screening.
16. Treatment with weight loss agents (e.g., orlistat, sibutramine, topiramate, bupropion) in the last 12 weeks prior to screening.
17. Treatment with mineral oil or fiber supplementation (e.g., Benefiber, Metamucil, among others).
18. Treatment with lipid-lowering drugs which have not been kept on a stable dose for the past 8 weeks before screening.
19. Treatment with thyroid replacement hormones which has not been kept on a stable dose for the past 12 weeks prior to screening.
20. Use of drugs under investigation within 30 days or 5 half-lives (whichever is longer) before screening unless the guidelines of local health authorities require a longer period.
21. Any of the following laboratory abnormalities identified in the screening by history and / or tests brought by the patient or that are part of this protocol, as described in section 4.3.4.6 of this project:

    21.1. Alanine aminotransferase (ALT) and / or Aspartate aminotransferase (AST) > 3 times the upper limit of normal 21.2. Glomerular filtration rate estimated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation ≤ 30 ml per min per 1,73 m2 21.3. Thyroid stimulating hormone (TSH) outside the normal range 21.4. Fasting triglycerides ≥ 400 mg / dL. 21.5. History of active substance abuse (including alcohol) within the past year
22. Any condition or concomitant medical disorder, not provided for in other items which in the opinion of the investigator, probably:

    22.1. Interfere with the patient's ability to complete the entire study period or participate in all activities of the study 22.2. Require during the study, administration of a treatment that may affect the interpretation of efficacy and safety data
23. Patients potentially unreliable and those considered by the investigator as unsuitable for the study

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-05 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 4 weeks
  3% weight loss

SECONDARY OUTCOMES:
Changes in hormone levels after 4 week treatment | baseline and 4 weeks
  Changes in hormone levels of satiety, appetite and endocrine pancreas, such as insulin comparing baseline to end of intervention.
Glycated Albumin | baseline and 4 weeks
  Reduction in fasting glycated albumin compared to baseline
Fasting Plasma Glucose | baseline and 4 weeks
  Reduction in fasting plasma glucose from baseline
Homeostatic Model Assessment (HOMA) | 4 weeks
  Insulin sensitivity index (HOMA-S) and Beta-cell dysfunction (HOMA-beta)
Body Mass Index (BMI) | 4 weeks
  Number of patients who achieved a BMI reduction unit
Intake of calories | 4 weeks
  Reduction or maintenance of the prescribed intake of calories during the 4-week intervention, in kcal/day, using a 3 days of food record, with food weighing.
Weight, waist circumference and total body fat loss after 3 and 6 month of end of intervention | 3 and 6 month after end of intervention
  weight and waist circumference loss

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Gerchman, MD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sumithran P, Prendergast LA, Delbridge E, Purcell K, Shulkes A, Kriketos A, Proietto J. Long-term persistence of hormonal adaptations to weight loss. N Engl J Med. 2011 Oct 27;365(17):1597-604. doi: 10.1056/NEJMoa1105816. PMID 22029981
- [Background] Schur EA, Kleinhans NM, Goldberg J, Buchwald D, Schwartz MW, Maravilla K. Activation in brain energy regulation and reward centers by food cues varies with choice of visual stimulus. Int J Obes (Lond). 2009 Jun;33(6):653-61. doi: 10.1038/ijo.2009.56. Epub 2009 Apr 14. PMID 19365394
- [Background] Boggio PS, Zaghi S, Villani AB, Fecteau S, Pascual-Leone A, Fregni F. Modulation of risk-taking in marijuana users by transcranial direct current stimulation (tDCS) of the dorsolateral prefrontal cortex (DLPFC). Drug Alcohol Depend. 2010 Dec 1;112(3):220-5. doi: 10.1016/j.drugalcdep.2010.06.019. Epub 2010 Aug 21. PMID 20729009
- [Background] Fregni F, Orsati F, Pedrosa W, Fecteau S, Tome FA, Nitsche MA, Mecca T, Macedo EC, Pascual-Leone A, Boggio PS. Transcranial direct current stimulation of the prefrontal cortex modulates the desire for specific foods. Appetite. 2008 Jul;51(1):34-41. doi: 10.1016/j.appet.2007.09.016. Epub 2007 Dec 23. PMID 18243412
- [Background] Goldman RL, Borckardt JJ, Frohman HA, O'Neil PM, Madan A, Campbell LK, Budak A, George MS. Prefrontal cortex transcranial direct current stimulation (tDCS) temporarily reduces food cravings and increases the self-reported ability to resist food in adults with frequent food craving. Appetite. 2011 Jun;56(3):741-6. doi: 10.1016/j.appet.2011.02.013. Epub 2011 Feb 23. PMID 21352881
- [Background] Montenegro RA, Okano AH, Cunha FA, Gurgel JL, Fontes EB, Farinatti PT. Prefrontal cortex transcranial direct current stimulation associated with aerobic exercise change aspects of appetite sensation in overweight adults. Appetite. 2012 Feb;58(1):333-8. doi: 10.1016/j.appet.2011.11.008. Epub 2011 Nov 12. PMID 22108669
- [Background] Kekic M, McClelland J, Campbell I, Nestler S, Rubia K, David AS, Schmidt U. The effects of prefrontal cortex transcranial direct current stimulation (tDCS) on food craving and temporal discounting in women with frequent food cravings. Appetite. 2014 Jul;78:55-62. doi: 10.1016/j.appet.2014.03.010. Epub 2014 Mar 20. PMID 24656950
- [Background] Lapenta OM, Sierve KD, de Macedo EC, Fregni F, Boggio PS. Transcranial direct current stimulation modulates ERP-indexed inhibitory control and reduces food consumption. Appetite. 2014 Dec;83:42-48. doi: 10.1016/j.appet.2014.08.005. Epub 2014 Aug 13. PMID 25128836
- [Background] Jauch-Chara K, Kistenmacher A, Herzog N, Schwarz M, Schweiger U, Oltmanns KM. Repetitive electric brain stimulation reduces food intake in humans. Am J Clin Nutr. 2014 Oct;100(4):1003-9. doi: 10.3945/ajcn.113.075481. Epub 2014 Aug 6. PMID 25099550
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Background] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Background] Brunoni AR, Nitsche MA, Bolognini N, Bikson M, Wagner T, Merabet L, Edwards DJ, Valero-Cabre A, Rotenberg A, Pascual-Leone A, Ferrucci R, Priori A, Boggio PS, Fregni F. Clinical research with transcranial direct current stimulation (tDCS): challenges and future directions. Brain Stimul. 2012 Jul;5(3):175-195. doi: 10.1016/j.brs.2011.03.002. Epub 2011 Apr 1. PMID 22037126
- [Background] Gandiga PC, Hummel FC, Cohen LG. Transcranial DC stimulation (tDCS): a tool for double-blind sham-controlled clinical studies in brain stimulation. Clin Neurophysiol. 2006 Apr;117(4):845-50. doi: 10.1016/j.clinph.2005.12.003. Epub 2006 Jan 19. PMID 16427357
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Bertolazi AN, Fagondes SC, Hoff LS, Pedro VD, Menna Barreto SS, Johns MW. Portuguese-language version of the Epworth sleepiness scale: validation for use in Brazil. J Bras Pneumol. 2009 Sep;35(9):877-83. doi: 10.1590/s1806-37132009000900009. English, Portuguese. PMID 19820814
- [Background] Graff SK, Alves BC, Toscani MK, Spritzer PM. Benefits of pedometer-measured habitual physical activity in healthy women. Appl Physiol Nutr Metab. 2012 Feb;37(1):149-56. doi: 10.1139/h11-145. Epub 2012 Jan 30. PMID 22288927
- [Background] Gorenstein C, Andrade L. Validation of a Portuguese version of the Beck Depression Inventory and the State-Trait Anxiety Inventory in Brazilian subjects. Braz J Med Biol Res. 1996 Apr;29(4):453-7. PMID 8736107
- [Background] Juraschek SP, Steffes MW, Miller ER 3rd, Selvin E. Alternative markers of hyperglycemia and risk of diabetes. Diabetes Care. 2012 Nov;35(11):2265-70. doi: 10.2337/dc12-0787. Epub 2012 Aug 8. PMID 22875225
- [Background] Liebetanz D, Koch R, Mayenfels S, Konig F, Paulus W, Nitsche MA. Safety limits of cathodal transcranial direct current stimulation in rats. Clin Neurophysiol. 2009 Jun;120(6):1161-7. doi: 10.1016/j.clinph.2009.01.022. Epub 2009 Apr 28. PMID 19403329
- [Derived] de Araujo C, Fitz RC, Natividade GR, Osorio AF, Merello PN, Schoffel AC, Brietzke E, Azevedo MJ, Schestatsky P, Gerchman F. The effect of transcranial direct current stimulation along with a hypocaloric diet on weight loss in excessive weight people: A pilot randomized clinical trial. Clin Nutr ESPEN. 2020 Dec;40:68-76. doi: 10.1016/j.clnesp.2020.10.005. Epub 2020 Oct 22. PMID 33183574
- [Derived] Araujo C, Fitz RC, Nogara DA, Schestatsky P, Gerchman F. Effect of transcranial direct current stimulation associated with hypocaloric diet on weight loss and metabolic profile in overweight or obesity: study protocol for a double-blind, randomized controlled clinical trial. Trials. 2018 Jul 16;19(1):386. doi: 10.1186/s13063-018-2776-3. PMID 30012180